CLINICAL TRIAL: NCT06454292
Title: Efficacy and Safety Study of Oliceridine Fumarate Versus Remifentanil for Analgesic Therapy in Mechanically Ventilated Subjects in the ICU
Brief Title: Efficacy and Safety Studies of Oliceridine Fumarate
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chun Pan (Other)
Responsible Party: Sponsor-Investigator, Chun Pan, professor, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-10
Record Dates: First submitted 2024-06-02; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group：Oliceridine Fumarate (Experimental)
  Interventions: Drug: Oliceridine Fumarate
- Control group: Remifentanil (Experimental)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Oliceridine Fumarate — After subjects were enrolled, the original sedative and analgesic drugs were discontinued, and a starting dose of 6ug/kg/h of oliceridine fumarate was continuously pumped, and the time of oliceridine fumarate initiation was recorded as T0. Subjects were assessed for sedation using the RASS score, and for analgesia using the CPOT score. Waiting for the original sedative-analgesic drug to elute until CPOT ≥ 3 and RASS > 0. Adjust the infusion rate of oliceridine fumarate according to the CPOT score (recommended to be adjusted by 2ug/kg/h, the range of adjustment is 2-20 ug /kg/h, and the maximum infusion rate is not more than 20 ug /kg/h) until the analgesic score of the subject is CPOT<3. The interval between two trial drug rate adjustments should be ≧5 min, and a CPOT score should be performed before each drug adjustment.
  Arms: Intervention group：Oliceridine Fumarate
Drug: Remifentanil — After subjects were enrolled, the original sedative and analgesic drugs were discontinued, and remifentanil was continuously pumped at a starting dose of 1.5ug/kg/h. The time of remifentanil initiation was recorded as T0. Subjects were assessed for sedation using the RASS score and analgesia using the CPOT score. We waited for the original sedative-analgesic drugs to elute until CPOT ≥ 3 and RASS > 0. The infusion rate of remifentanil was adjusted according to the CPOT score (1.5ug/kg/h is recommended, the range of adjustment is 1.5~12μg/kg/h, and the maximum infusion rate is not more than 12μg/kg/h) until the subject's analgesic score of CPOT<3, and the interval between the two experimental rate adjustments of the drug should be ≧5min, and the CPOT score should be performed before each adjustment of the drug. The CPOT score should be performed before each drug adjustment.
  Arms: Control group: Remifentanil

SUMMARY:
The objective of this clinical trial is to investigate the efficacy and safety of oliceridine fumarate for analgesic treatment in mechanically ventilated subjects in the ICU. This study was conducted to answer the following questions (1) the efficacy of oliceridine fumarate for analgesic treatment in subjects with ICU mechanical ventilation (2) the safety of oliceridine fumarate for analgesic treatment in subjects with ICU mechanical ventilation. This study proposes to conduct a randomized controlled clinical trial in mechanically ventilated patients in the intensive care unit to compare the analgesic efficacy and incidence of adverse effects of two drugs, oliceridine fumarate injection and remifentanil. Subjects had an analgesic goal of CPOT <3 points and a sedation goal of RASS -2 to 0 points. Infusion syringes of remifentanil or oliceridine fumarate were prepared by a nurse according to the weight of the subjects. Subjects were enrolled in the group and were scored for analgesia and sedation related scores. Both groups received routine ICU monitoring and appropriate treatment, which was determined by the clinician.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years and ≤80 years;
2. Admitted to the ICU and undergoing invasive mechanical ventilation with an expected duration of mechanical ventilation of more than 24 hours;
3. Subjects requiring sedation and analgesia;
4. Subjects or their guardians voluntarily participate in the study and sign an informed consent form;

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. Hypersensitivity to opioids (fentanyl, remifentanil, sufentanil, morphine, etc.);
3. Subjects with bronchial asthma attacks;
4. Subjects with acute intestinal obstruction;
5. Subjects who are unable to undergo RASS and CPOT assessments for various reasons, such as those with a history of psychiatric systemic disorders (schizophrenia, mania, psychosis, history of cognitive dysfunction), grand mal status epilepticus, and craniocerebral injury;
6. Severe hemodynamic instability (subjects who require administration of more than an equivalent dose of 0.5 μg/kg/min norepinephrine to maintain a MAP ≥ 65 mmHg and who, in the opinion of the investigator, are not suitable for enrollment);
7. Use of monooxygenase inhibitors (MAOIs) (see protocol appendix);
8. Chronic pain requiring long-term analgesic medication (duration of illness greater than 3 months);
9. Severe hepatic insufficiency (liver function in Child classification C);
10. Severe renal dysfunction (definition of renal dysfunction: chronic renal insufficiency [glomerular filtration rate (GFR) ≦29ml/(min1.73m3]; or long-term maintenance hemodialysis or peritoneal dialysis subjects);
11. Undergoing any clinical trial within 1 month prior to enrollment and receiving the test product;
12. ECG QT interval at screening: >450 ms for men and >470 ms for women;
13. Subjects with a desired sedation target RASS score within the range of -5 to -3 (including threshold) points;
14. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of analgesic effectiveness | Not more than 3 days
  Percentage of time to achieve analgesic goal as a percentage of total time on medication during the study drug efficacy period (analgesic goal was CPOT <3 points, and the start of recording was the time of initiation of medication).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo JC, Lu S, Fu XL, Shen J, He HL, Pan C, Huang XB. Comparison of Oliceridine to Remifentanil for Optimal Analgesia in Mechanical Ventilation (CO-ROAM): Study Protocol for a Multicenter Randomized Controlled Trial. Pain Ther. 2024 Dec;13(6):1695-1704. doi: 10.1007/s40122-024-00669-4. Epub 2024 Oct 18. PMID 39424775